CLINICAL TRIAL: NCT00130195
Title: Phase 2 Study of Imatinib-Combined Chemotherapy for Newly Diagnosed BCR-ABL-Positive Acute Lymphoblastic Leukemia
Brief Title: Study of Imatinib-Combined Chemotherapy for BCR-ABL-Positive Acute Lymphoblastic Leukemia (ALL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Japan Adult Leukemia Study Group (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JALSG Ph+ALL202
Record Dates: First submitted 2005-08-12; First posted 2005-08-15 (Estimated); Last update posted 2008-11-14 (Estimated); Status verified 2008-11

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: acute lymphoblastic leukemia; BCR-ABL; Philadelphia-chromosome; newly diagnosed
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Philadelphia Chromosome | interventions — Imatinib Mesylate; Cyclophosphamide; Daunorubicin; Vincristine; Prednisolone; Methotrexate; Cytarabine; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Drug: imatinib; Drug: cyclophosphamide; Drug: daunorubicin; Drug: vincristine; Drug: prednisolone; Drug: methotrexate; Drug: cytarabine; Drug: dexamethasone

INTERVENTIONS:
Drug: imatinib
Drug: cyclophosphamide
Drug: daunorubicin
Drug: vincristine
Drug: prednisolone
Drug: methotrexate
Drug: cytarabine
Drug: dexamethasone

SUMMARY:
The purpose of this study is to determine the clinical efficacy and safety of imatinib-combined chemotherapy on newly diagnosed BCR-ABL-positive ALL.

DETAILED DESCRIPTION:
Philadelphia chromosome (Ph) is a translocation abnormality leading to the formation of the BCR-ABL gene rearrangement. This genetic abnormality occurs in up to 30% of adult acute lymphoblastic leukemia (ALL), and its presence is known to be the most adverse prognostic factor for ALL. Because long-term survival cannot be achieved by conventional chemotherapy alone, there is a clear medical need for alternative treatment approaches. Imatinib is a potent selective inhibitor of the BCR-ABL protein kinase, and it has been reported that single-agent imatinib induced response in a substantial proportion of Ph-positive ALL (Ph+ALL) patients, but that the response was not durable. The Japan Adult Leukemia Study Group (JALSG) has therefore started a phase 2 study designed to evaluate the clinical effect of imatinib-combined chemotherapy on newly diagnosed BCR-ABL-positive ALL.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated BCR-ABL-positive ALL
* Age between 15 and 64 years
* Performance status between 0 and 3 (ECOG criteria)
* Adequate functioning of the liver (serum bilirubin level < 2.0 mg/dL), kidneys (serum creatinine level < 2.0 mg/dL), and heart (left ventricular ejection fraction greater than 50% and no severe abnormalities detected on electrocardiograms and echocardiographs)
* Written informed consent to participate in the trial

Exclusion Criteria:

* Uncontrolled active infection
* Another severe and/or life-threatening disease
* Positive for HIV antibody and/or hepatitis B surface (HBs) antigen tests
* Another primary malignancy which is clinically active and/or requires medical interventions
* Pregnant and/or lactating women
* Past history of renal failure

Ages: 15 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2002-09; Primary Completion 2008-02 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The rate of complete remission | 63 days

SECONDARY OUTCOMES:
The duration of remission | 1 year
Overall survival | 1 year
Toxicity caused by combination of imatinib and chemotherapy | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Fumihiko Hayakawa, MD, Study Director — Nagoya University; Tomoki Naoe, MD, Study Chair — Nagoya University
Locations (1):
- Department of Hematology, Nagoya University Graduate School of Medicine, Nagoya, Japan

REFERENCES:
- [Result] Towatari M, Yanada M, Usui N, Takeuchi J, Sugiura I, Takeuchi M, Yagasaki F, Kawai Y, Miyawaki S, Ohtake S, Jinnai I, Matsuo K, Naoe T, Ohno R; Japan Adult Leukemia Study Group. Combination of intensive chemotherapy and imatinib can rapidly induce high-quality complete remission for a majority of patients with newly diagnosed BCR-ABL-positive acute lymphoblastic leukemia. Blood. 2004 Dec 1;104(12):3507-12. doi: 10.1182/blood-2004-04-1389. Epub 2004 Aug 17. PMID 15315963
- [Result] Yanada M, Takeuchi J, Sugiura I, Akiyama H, Usui N, Yagasaki F, Kobayashi T, Ueda Y, Takeuchi M, Miyawaki S, Maruta A, Emi N, Miyazaki Y, Ohtake S, Jinnai I, Matsuo K, Naoe T, Ohno R; Japan Adult Leukemia Study Group. High complete remission rate and promising outcome by combination of imatinib and chemotherapy for newly diagnosed BCR-ABL-positive acute lymphoblastic leukemia: a phase II study by the Japan Adult Leukemia Study Group. J Clin Oncol. 2006 Jan 20;24(3):460-6. doi: 10.1200/JCO.2005.03.2177. Epub 2005 Dec 12. PMID 16344315
- [Result] Yanada M, Takeuchi J, Sugiura I, Akiyama H, Usui N, Yagasaki F, Nishii K, Ueda Y, Takeuchi M, Miyawaki S, Maruta A, Narimatsu H, Miyazaki Y, Ohtake S, Jinnai I, Matsuo K, Naoe T, Ohno R; Japan Adult Leukemia Study Group. Karyotype at diagnosis is the major prognostic factor predicting relapse-free survival for patients with Philadelphia chromosome-positive acute lymphoblastic leukemia treated with imatinib-combined chemotherapy. Haematologica. 2008 Feb;93(2):287-90. doi: 10.3324/haematol.11891. Epub 2008 Jan 26. PMID 18223280
- See also: The JALSG homepage — http://www.jalsg.jp/